CLINICAL TRIAL: NCT06388915
Title: A Retrospective Cohort Study of 15 Cases of Pelvic Fractures Complicated by Morel-Lavallee Lesion
Status: Completed | Type: Observational
Sponsor: Weikang Chen (Other)
Responsible Party: Sponsor-Investigator, Weikang Chen, Graduate student in bone surgery, Fujian Provincial Hospital
Organization: Fujian Provincial Hospital (Other)
Other Study IDs: K2202403004
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Pelvic Fracture; Morel-Lavallee Lesion
Keywords: Morel-Lavallee Lesion; Pelvic Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Some related factors of pelvic fracture and Morel-Lavallee injury (MLL) are preliminarily discussed, which provides some preliminary references for early clinical detection and research of such injuries.

DETAILED DESCRIPTION:
Inclusion criteria: (1) The clinical symptoms are consistent with the diagnosis of pelvic fracture, and the diagnosis is confirmed by imaging, including emergency or sub-emergency CT data within 72 hours after injury. (2) The symptoms of the diagnosis of MLL were pain and swelling at the site of occurrence, a sense of soft tissue fluctuation found on physical examination, and a complete process of puncture drainage + negative pressure suction therapy. (3) The patients and their families have given informed consent to this study and signed the informed consent form, which meets the ethical requirements.

Exclusion criteria: (1) Incomplete imaging data, especially the lack of emergency or sub-emergency CT data within 72 hours after injury. (2) Cases of other severe lower limb fractures such as femur and trochanter, and lower limb fractures combined with MLL injury have been reported in the literature.

ELIGIBILITY:
Inclusion Criteria:

* (1) The clinical symptoms are consistent with the diagnosis of pelvic fracture, and the diagnosis is confirmed by imaging, including emergency or sub-emergency CT data within 72 hours after injury. (2) The symptoms of the diagnosis of MLL were pain and swelling at the site of occurrence, a sense of soft tissue fluctuation found on physical examination, and a complete process of puncture drainage + negative pressure suction therapy. (3) The patients and their families have given informed consent to this study and signed the informed consent form, which meets the ethical requirements.

Exclusion Criteria:

* (1) Incomplete imaging data, especially the lack of emergency or sub-emergency CT data within 72 hours after injury. (2) Cases of other severe lower limb fractures such as femur and trochanter, and lower limb fractures combined with MLL injury have been reported in the literature.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 206 cases of pelvic fractures, including 15 cases with MLL complications, were collected between June 2017 and June 2023.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-23 (Actual)

PRIMARY OUTCOMES:
Site of MLL | 5 days
  Site of the occurrence of Morel-Lavallee lesion
Site of injury and Classification of pelvic fracture | 72 hours
  Site of injury and Classification of pelvic fracture

SECONDARY OUTCOMES:
Time to treatment | 10 days
  Time of treatment for Morel-Lavallee lesion
Drainage volume | 10 days
  Drainage volume for Morel-Lavallee lesion

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No